CLINICAL TRIAL: NCT05359718
Title: The Psychological Impact of COVID-19 on Patients with Solid Malignancies: a Single-Institution Survey Study
Acronym: PICO SM
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp196
Record Dates: First submitted 2021-03-08; First posted 2022-05-04 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
The COVID-19 pandemic and the subsequent government-imposed restrictions have undeniably resulted in unprecedented changes to the life of patients with cancer. It has become more evident that patients with cancer may be at significant risk of higher morbidity and mortality when infected with SARS-CoV-2, which is understandably causing anxiety amongst both patients and their oncology team.

This project is a single centre, non-interventional observational prospective cohort study; which aims to evaluate the impact of COVID-19 on the mental health and general wellbeing of patients diagnosed with solid malignancies by utilising a range of non-invasive questionnaires (GAD-7, PHQ-9, PC-PTSD-5, WHO-5 and Wellbeing thermometer). Data on patient demographics, treatment and medical history, and medical resource utilization will be obtained through a medical chart review at enrolment for up to 4 months. Participants will be asked to complete five questionnaires regarding their mental health and wellbeing status during their routine clinic visits, but no other additional tests or procedures will be undertaken for the study outside of their routine care.

It is essential to understand both the short and long term psychological consequences of COVID-19 on cancer patients to better inform the institute and other regional and national stakeholders of the scale of the issue, in order to recommend necessary measures and resources required to address this important issue.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or over.
2. Cancer diagnosis
3. Able to fully comprehend the Patient Information Sheet

Exclusion Criteria:

1. Patients who lack capacity to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the levels of anxiety, depression, post-traumatic stress and well-being amongst patients with cancer during the COVID-19 pandemic using Generalised Anxiety Disorder Assessment (GAD-7) | 12 months
  Psychometric Measure - higher scores indicates greater anxiety
To evaluate the levels of anxiety, depression, post-traumatic stress and well-being amongst patients with cancer during the COVID-19 pandemic using PHQ-9 (Patient Health Questionnaire-9) | 12 months
  Psychometric Measure, higher score indicates greater depression
To evaluate the levels of anxiety, depression, post-traumatic stress and well-being amongst patients with cancer during the COVID-19 pandemic using The Primary Care Post-Traumatic Stress Disorder (PC-PTSD-5) | 12 months
  Psychometric Measure, higher scores indicates greater risk of Post-Traumatic Stress Disorder
To evaluate the levels of anxiety, depression, post-traumatic stress and well-being amongst patients with cancer during the COVID-19 pandemic using World Health Organisation Five-Wellbeing Index | 12 months
  Psychometric Measure, assesses general psychological wellbeing
To evaluate the levels of anxiety, depression, post-traumatic stress and well-being amongst patients with cancer during the COVID-19 pandemic using Well-being thermometer | 12 months
  Psychometric Measure

SECONDARY OUTCOMES:
To determine the factors contributing to anxiety, depression and post-traumatic stress during COVID-19 determined by the above questionnaires | 12 months
  GAD-7
To determine the factors contributing to anxiety, depression and post-traumatic stress during COVID-19 determined by the above questionnaires | 12 months
  PHQ-9
To determine the factors contributing to anxiety, depression and post-traumatic stress during COVID-19 determined by the above questionnaires | 12 months
  PC-PTSD-5
To understand the needs of cancer patients during the period of a pandemic in order to help further develop immediate and longer term support measures | 12 months
  By assessing WHO-5
To understand the needs of cancer patients during the period of a pandemic in order to help further develop immediate and longer term support measures | 12 months
  By assessing thermometer questionnaires.
To correlate the novel well-being thermometer with existing psychometric scales as a screening tool for future patient assessment. | 12 months
  Correlating the Well-being thermometer with the above psychometric measures.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No